CLINICAL TRIAL: NCT00686933
Title: The Long-Term Safety and Tolerability of ABT-089 in Adults With Attention Deficit-Hyperactivity Disorder (ADHD): An Open-Label Extension Study for Subjects Completing Study M10-346
Brief Title: Long Term Safety and Tolerability Study of ABT-089 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-425
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pozanicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-089

INTERVENTIONS:
Drug: ABT-089 — Subjects will take up to 80 mg daily for 24 months

SUMMARY:
The objective of this study is to evaluate the long-term effects and tolerability of ABT-089 in adults with Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* The subject was randomized into Study M10-346 and completed the study.
* Female subjects of childbearing potential must have a negative urine pregnancy test at screening and baseline and agree to comply with applicable contraceptive requirements.
* Male subjects must agree to comply with applicable contraceptive requirements.
* The subject is judged to be in generally good health.

Exclusion Criteria:

* The subject has taken any ADHD medication between the last dose of study drug in Study M10-346 and the first dose of study drug in the current study.
* The subject anticipates a move outside the geographic area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
CAARS:Inv | Day -1, Day 14, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24
CGI-ADHD-S | Day -1, Day 14, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24

SECONDARY OUTCOMES:
CAARS:Self | Day -1, Day 14, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24
BRIEF-A | Day -1, Month 3, 6, 9, 12, 15, 18, 21, 24
AAQOL | Day -1, Month 3, 6, 9, 12, 15, 18, 21, 24
WPAI | Day -1, Month 3, 6, 9, 12, 15, 18, 21, 24
FTND | Day -1, Month 1, 2, 3, 6, 9, 12, 15, 18, 21, 24

CONTACTS AND LOCATIONS:
Overall Officials: Earle Bain, MD, Study Director — AbbVie
Locations (12):
- United States (12):
  - Site Reference ID/Investigator# 8315, Lafayette, California
  - Site Reference ID/Investigator# 8306, Jacksonville, Florida
  - Site Reference ID/Investigator# 8308, Orlando, Florida
  - Site Reference ID/Investigator# 8314, Overland Park, Kansas
  - Site Reference ID/Investigator# 8307, Farmington Hills, Michigan
  - Site Reference ID/Investigator# 8318, Troy, Michigan
  - Site Reference ID/Investigator# 8309, Eugene, Oregon
  - Site Reference ID/Investigator# 8316, Portland, Oregon
  - Site Reference ID/Investigator# 8310, Memphis, Tennessee
  - Site Reference ID/Investigator# 8319, Virginia Beach, Virginia
  - Site Reference ID/Investigator# 8305, Bellevue, Washington
  - Site Reference ID/Investigator# 8320, Seattle, Washington